CLINICAL TRIAL: NCT06529536
Title: Genotype Informed Bayesian Dosing of Tacrolimus in Solid Organ Transplant- Pharmacogenomic Implementation in Children
Brief Title: Utilising Genotype Informed Bayesian Dosing of Tacrolimus in Children Post Solid Organ Transplantation.
Acronym: BRUNO-PIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/ETH02699
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Solid Organ Transplant
Keywords: Tacrolimus; Pharmacogenomics; Bayesian; Paediatrics
MeSH Terms: interventions — Genotype; Tacrolimus

STUDY DESIGN:
Intervention Model Description: This is an open-label trial with a prospective intervention arm and a retrospective standard of care comparator arm. Forty-five SOT recipients will be recruited from The Royal Children's Hospital Melbourne (with retrospective controls taken from the immediately prior 5 years).
  For all eligible SOT patients, a pre-emptive CYP3A5 and CYP3A4 genotype will be combined with a population PK model to predict optimal initial tacrolimus dose. In addition, genotype-informed Bayesian revised dosing will be applied to all transplant recipients over the subsequent 8-weeks post-transplant.
  The prospective arm will be compared with a retrospective arm (using standard mg/kg dosing plus therapeutic drug monitoring) where the primary outcome is the proportion of each cohort with tacrolimus concentration (steady-state average concentration) within the acceptable range of 80-125% of target at post-transplant dosing day 4 (DD4), at week 3 and at week 8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prospective Cohort: Pre-emptive CYP3A5/3A4 genotype combined with a Bayesian dose prediction (Experimental): Planned SOT recipients where initial tacrolimus dosing will be based on genotype and subsequent doses predicted using Bayesian revised dosing using NextDose. NextDose, a web-based tool is a model-informed precision dosing software tool used to optimise dosage regimens. It uses Bayesian statistics to integrate prior drug information from a population pharmacokinetic (popPK) model, individual characteristics, and drug concentrations to provide the most accurate individual pharmacokinetic (PK) estimates. The popPK model, a mathematical-statistical model developed from real patient data, captures the drug's typical pharmacokinetics, its variability among individuals and over time, and the factors influencing this variability. By leveraging prior knowledge about a drug's PK along with individual patient data and drug concentrations, the software accurately estimates individual PK parameters with minimal drug concentration data. Tacrolimus dose, form, frequency, & duration will be assessed
  Interventions: Diagnostic Test: Genotyping for CYP3A4 and CYP3A5 genes; Device: Use of NextDose platform; Drug: Tacrolimus

INTERVENTIONS:
Diagnostic Test: Genotyping for CYP3A4 and CYP3A5 genes — Genotyping: Patients in the prospective (intervention) arm will undergo genotyping using Illumina's genome-wide genotyping array (Infinium Global Screening Array). Pre-transplant genotyping will test for CYP3A5 *3, *6, *7, *8 and *9 alleles, and will test for CYP3A4*22 only (with CYP3A4*1 reported if no variant corresponding to *22 was present).
  The determined diplotypes for CYP3A5 will be matched with predicted phenotypes using the Clinical Pharmacogenetics Implementation Consortium (CPIC®) proposed genotype-to-phenotype translation table. The assignment of the phenotype is outlined in the CPIC guidelines which will used to predict initial dose of tacrolimus. In addition, influence of CYP3A4 will be incorporated based on recent literature and interventional trials. Initial dose in BRUNO-PIC will use allometric size scaling from adult dose, with adjustment based on genotype (CYP3A4 & CYP3A5)
Device: Use of NextDose platform — NextDose platform is a forecasting tool used to predict tacrolimus dosage. It is a freely available tool and will be used in accordance with guideline. The dosing recommendations will be led by the academic pharmacist in consultation with the PI. This tool will use genotype-informed Bayesian dosing to help predict the time course of tacrolimus concentrations in the body.
Drug: Tacrolimus — Tacrolimus is administered to all patients post SOT at The Royal Children's Hospital (RCH)
  Other Names: Prograf (Brand)

SUMMARY:
This study aims to evaluate the efficacy of genotype-informed Bayesian dosing of tacrolimus in optimising drug exposure among paediatric solid organ transplant recipients. By tailoring tacrolimus dosage based on individual genetic makeup and using Bayesian modeling to predict drug levels, the researchers hope to increase the likelihood of achieving therapeutic drug concentrations while minimising the risk of adverse events associated with subtherapeutic or supratherapeutic exposure.

DETAILED DESCRIPTION:
Tacrolimus, a calcineurin inhibitor is an effective immunosuppressant for solid organ transplants (SOT). Due to its narrow therapeutic index and individual variability in its pharmacokinetics (PK), this can lead to inefficacy, toxicities and suboptimal outcomes.

Tacrolimus is typically administered orally twice daily, with a starting dose scaled linearly to body weight (mg/kg). Dose is then adjusted based on measured steady-state trough (pre-dose) whole blood tacrolimus concentrations, to bring to within a desired "therapeutic range". However, this dosing strategy remains associated with incomplete effectiveness and toxicities in a substantial proportion of recipients, related to under- or over-exposure respectively.

Cytochrome P450 CYP3A4 and CYP3A5 enzymes metabolise tacrolimus, with research suggesting a link between the CYP3A5 genetic makeup and achieving tacrolimus target levels. Genotyping for the CYP3A5 gene prior to SOT can identify individuals who are at risk of high or low tacrolimus levels, and guide tacrolimus dosing prior to transplantation. Bayesian prediction is a pharmaco-statistical technique that uses population pharmacokinetic data and individual patient characteristics to accurately predict the tacrolimus dose required to achieve a target concentration. Subtherapeutic levels post-transplant, increases the risk of acute rejection. Furthermore, failure to maintain the target tacrolimus range for the first 6 months significantly raises the chance of rejection, donor-specific antibody formation and graft loss.

Genotype informed dosing algorithms may optimise and ameliorate sub-therapeutic levels, thus potentially reducing the risk of rejection or toxicity.

To determine if implementing a genotype-informed Bayesian dosing of tacrolimus is superior to standard weight-based dosing and empiric dose adjustment to trough concentrations post SOT, a combined retrospective/prospective cohort study in Solid Organ Transplant recipients will be undertaken at The Royal Children's Hospital Melbourne.

The outcomes from the Retrospective cohort (over a 5-year period) using clinician-led therapeutic drug monitoring will be compared with the Prospective cohort (n=45), using genotype to predict initial tacrolimus doses and predictive Bayesian dosing for ongoing tacrolimus dosing over a 8-week period.

ELIGIBILITY:
Participants will be assigned to the prospective arm if treated at Royal Children's Hospital who are receiving a solid organ transplant (SOT) (excluding repeat graft in liver transplant recipients) and who will be on tacrolimus as one of the main immunosuppressants post-transplant.

Inclusion Criteria:

* 1 to 18years old
* SOT transplant (planned or on waiting list).
* Heart OR Liver OR Renal transplant recipients
* Amenable to venepuncture and blood draw
* Patient and/or parent consented to the study.

Exclusion Criteria:

* older than 18 year old
* younger than 1 year old
* Previous liver transplant.
* Lung OR Intestinal transplant.
* Insufficient time before transplant for pharmacogenomic analysis (prospective arm only)
* Patient has a known hypersensitivity to tacrolimus and/or its formulation.
* On a slow release preparation of Tacrolimus (e.g Advagraf extended release Brand)
* Immunosuppressant regimen not containing tacrolimus immediate release product
* Patient and/or parent is unable to consent to the study.
* Patient and/or parent is unwilling to take part in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Proportion of cohort with tacrolimus concentration within 80-125% of concentration target (Cssavg: average steady state concentration) on post-transplant dosing day 4 (DD4), Week 3 and Week 8 | Post transplantation at Day 4, Week 3 and week 8
  To measure the proportion of cohort with tacrolimus concentration within 80-125% of concentration target on post-transplant dosing day 4 (DD4), week 3 and week 8 - within 80-125% of Cssavg target (where Cssavg (average steady state concentration) is calculated using Bayesian maximum a posteriori estimation, from observed concentrations and clinical covariates)

SECONDARY OUTCOMES:
Proportion of cohort reaching acceptable concentrations. | Post transplantation through first 8-week period
  To measure the median time to acceptable range (80-125% Cssavg, steady state concentration) in the immediate post-transplant period.
Change in proportion of cohort to stay within acceptable range post-transplant period. | Post transplantation through first 8-week period
  To measure the time within acceptable range(80-125% of Cssavg, steady state concentration) in the first 8-weeks post-transplant
Change in proportion of cohort to stay within acceptable range immediately post-transplant. | Post transplantation at Day 4
  To measure the proportion of tacrolimus concentrations within 80-125% of Csstrough (steady state concentration) target on DD4
Number of dose adjustments of tacrolimus dosing post-transplantation | Post transplantation at Week 8
  To measure the number of dose adjustments of tacrolimus based on Therapeutic Drug Monitoring and/or Bayesian modelling.
Number of related adverse events in participants relating to using genotype-informed Bayesian dosing within the first 8 weeks post transplant | From first dose of Tacrolimus through to 8 weeks post transplantation
  To record any adverse events that occur relating to using genotyping and Bayesian dosing for dose prediction of tacrolimus. These include any subtherapeutic or supratherapeutic tacrolimus levels as a direct result of genotyping or Bayesian prediction.
Number of barriers in implementing genotype-informed Bayesian dosing | From first dose of Tacrolimus through to 8 weeks post transplantation
  To record any barriers that occur in using genotyping and Bayesian dosing for dose prediction of tacrolimus. These can include any technical failures of the NextDose platform for dosing predictions or data access.
Number of unfavorable clinical outcomes | From first dose of Tacrolimus to 8 weeks post transplantation
  To compare of the number of unfavorable clinical outcomes: rejection, donor-specific antibody formation and toxicities between the two cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Conyers, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of this study will be available six months after publication of the primary outcome. The study protocol and analysis plan will also be available. The data must be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the Study Management Group must see and approve the data analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the Study Management Group be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research organisation which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1. Data access agreement;
  2. approval by Trial Steering Committee;
  3. recognized research institutions.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre